CLINICAL TRIAL: NCT05383456
Title: The Visceral Adiposity Measurement and Observation Study
Acronym: VAMOS
Status: Completed | Type: Observational
Sponsor: Theratechnologies (Industry)
Collaborators: Dacima Consulting (Other); Medpace, Inc. (Industry); Vanderbilt University Medical Center (Other); Echosens (Industry)
Responsible Party: Sponsor
Other Study IDs: TH9507-CTR-1030
Record Dates: First submitted 2022-04-08; First posted 2022-05-20 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: HIV; HIV-Infections; HIV-1-infection; HIV I Infection; HIV Lipodystrophy; HIV Infection Primary; HIV-Associated Lipodystrophy; HIV Disease Progression; Lipohypertrophy; Liver Diseases; NAFLD; NASH; Liver Fibrosis; Hepatic Fibrosis; Waist Circumference; BMI; Ectopic Fat; Liver Fat; Hepatic Steatosis
Keywords: HIV; HIV Infections; HIV-1-infection; HIV Lipodystrophy; HIV Infection Primary; HIV-Associated Lipodystrophy; HIV Disease Progression; Lipohypertrophy; Liver Disease; NAFLD, Liver Fat, Hepatic Steatosis; NASH; Liver Fibrosis and Hepatic Fibrosis; Ectopic Fat; Pericardial Fat; Muscle Fat/Density; Liver CAP; Liver VTCE; Waist Circumference; Anthropometric Measurements; BMI; Hip Circumference; Waist to Hip Ratio
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV-Associated Lipodystrophy Syndrome; Liver Diseases; Non-alcoholic Fatty Liver Disease; Liver Cirrhosis; Fatty Liver; HIV Infections | interventions — Diagnostic Tests, Routine; Tomography, X-Ray Computed; Urination; Hematologic Tests

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum sample for lipid analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Participants: Waist and hip circumferences, CT Scan and FibroScan and Quality of Life questionnaire, vital signs, urine and blood testing in Adults with HIV on continuous Anti-Retroviral Therapy treatment.
  Interventions: Diagnostic Test: Diagnostic Test; Drug: HIV Anti-retroviral Background Therapy

INTERVENTIONS:
Diagnostic Test: Diagnostic Test — Standard diagnostic tests.
  Other Names: CT Scan; Fibroscan; Urine and Blood testing
Drug: HIV Anti-retroviral Background Therapy — All participants are required be on continuous HIV Anti-retroviral Background Therapy.
  No intervention on drug is part of the Study.

SUMMARY:
The Visceral Adiposity Measurement and Observation Study

DETAILED DESCRIPTION:
Visceral adiposity (VA) is a form of ectopic fat deposition that correlates with cardiometabolic risk in both the general population and among people with human immunodeficiency virus (HIV) (PWH).1 Excess VA (EVA) is prevalent among PWH,2,3 and prevalence rises with age and time on antiretroviral treatment.3 Effective plasma virologic suppression is not protective against EVA and associated comorbidities, possibly due to adverse metabolic effects of certain antiretroviral agents, the low-level expression of HIV gene products within the adipose tissue, and other factos.4

Although EVA has been reported to occur in nearly half of PWH on antiretroviral therapy (ART),2,3 it may go unrecognized or be mischaracterized as generalized obesity. Whereas obesity and EVA both increase waist circumference (WC), they differ in that overweight and obese individuals accumulate fat primarily in subcutaneous depots, whereas individuals with EVA accumulate fat within the abdominal cavity. Ectopic fat accumulation (EFA) also occurs at various other depots, namely around and within various internal organs (e.g., the heart, skeletal muscle, liver, and pancreas).1,5 For purposes of the VAMOS study, EFA is defined as the amount of pericardial fat, skeletal muscle fat, and liver fat the VAMOS study subjects have. VA for the VAMOS study is held separately as it is the primary endpoint.

Because it represents a potentially modifiable cardiovascular risk factor among PWH, simple, practical surrogate markers are needed to identify patients with probable EVA. Anthropometric measurements such as WC correlate with EVA in the general population1, but their predictive value is less well defined for subgroups of PWH.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, ≥18 years
2. HIV+, on continuous ART for ≥12 months
3. ≥3 years since initiation of ART
4. 20.0 ≤ BMI ≤ 40.0 kg/m2

Exclusion Criteria:

1. Detectable HIV plasma viremia 12 months prior enrollment, defined by ≥1 measurement of HIV-1 ribonucleic acid (RNA) > 1000/mL
2. Unable or unwilling to undergo any study procedures
3. Known hepatic cirrhosis
4. Active hepatitis C within past 12 months, defined by detectable hepatitis C RNA
5. Hepatitis B positive
6. Current pregnancy or breastfeeding
7. History of liver transplant
8. Self-reported weekly alcohol consumption meets National Institute on Alcohol Abuse and Alcoholism (NIAAA) criteria for problematic drinking (binge or chronic daily intake)
9. Any active malignancy, excluding non-melanoma skin cancer
10. Patient has been treated with tesamorelin or human growth hormone within the last 12 months
11. Patient has used insulin in the previous year
12. Patient has undergone bariatric surgery in the year prior to enrollment or is currently undergoing a weight loss program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Sex will be defined by sex assigned at birth.
  Gender will be by self-declared gender identity. Thus:
  * Men will include cis-identified males and trans men.
  * Women will include cis-identified women and trans women.
Study Population: The overall study population will include all participants who provide informed consent, are enrolled in the study, and complete all study procedures as required.
  The cardiovascular risk analysis population will not include participants who have history of CVD (myocardial infarction, cerebrovascular accident, heart failure, or atrial fibrillation).
  Diagnosis of normal versus excess VA using published criteria12,15,16,20 (normal visceral adiposity (NVA) versus EVA) will be based on CT evidence of VA cross-sectional area (<130cm2 or ≥130cm2, respectively).
Sampling Method: Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2022-04-18 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Umbilical waist circumference measurement (in cm). | Baseline
  Two types of waist circumference (WC) measurements (umbilical and iliac) will be assessed for a predicting relationship to Excess Visceral Adiposity (EVA) as measured by CT surface area.
Iliac waist circumference measurement (in cm). | Baseline
  Two types of waist circumference (WC) measurements (umbilical and iliac) will be assessed for a predicting relationship to Excess Visceral Adiposity (EVA) as measured by CT surface area.
Visceral Adiposity Measurement by CT surface area (cm2). | Baseline
  Two types of waist circumference (WC) measurements (umbilical and iliac) will be assessed for a predicting relationship to Excess Visceral Adiposity (EVA) as measured by CT surface area.

SECONDARY OUTCOMES:
Visceral Adiposity Measurement by CT surface area (cm2) | Baseline
  Two types of waist circumference (WC) measurements (Outcome 1 and Outcome 2) and BMI (Outcome 6) will be assessed for a predicting relationship to Excess Visceral Adiposity (EVA) as measured by CT surface area.
Visceral Adiposity Measurement by CT volume (cm3). | Baseline
  Two types of waist circumference (WC) measurements (Outcome 1 and Outcome 2) will be assessed for a relationship to Visceral Adiposity as measured by CT volume.
Weight in kg and height in meter will be combined to report body mass index (BMI) in kg/m2. | Baseline
  Two types of waist circumference (WC) measurements (Outcome 1 and Outcome 2) and BMI will be assessed for a predicting relationship to Visceral Adiposity as measured by CT surface area (Outcome 4), Visceral Adiposity as measured by CT volume (Outcome 5), Framingham Cardiovascular Risk strata (Outcome 9), Liver disease (Outcome 10 and 11) or Glucose homeostasis (Outcome 12).
Health related quality of life evaluation by SF-36 questionnaire | Baseline
  Quality of life will be assessed for a relationship to Visceral Adiposity as measured by CT surface area.
Health related quality of life evaluation by VAMOS disease specific questionnaire | Baseline
  Quality of life will be assessed for a relationship to Visceral Adiposity as measured by CT surface area.
Framingham Cardiovascular Risk strata (low, intermediate or high) | Baseline
  Participant age in year, HDL-cholesterol in mmol/L, Total Cholesterol in mmol/L and systolic blood pressure in mmHg will be combined to determine the Framingham Cardiovascular Risk strata (low, intermediate or high). Two types of waist circumference (WC) measurements (Outcome 1 and Outcome 2) will be assessed for a relationship to Framingham Cardiovascular Risk strata.
Fibroscan Controlled Attenuation Parameter (CAP) in decibels/minute | Baseline
  To evaluate liver disease (hepatic steatosis (HS))
Fibroscan Vibration Controlled Transient Elastography (VCTE) in kPa | Baseline
  To evaluate liver disease (hepatic fibrosis (HF))
Glucose homeostasis as measured by percentage (%) of glycated form of hemoglobin in blood (HbA1c). | Baseline
  Two types of waist circumference (WC) measurements (Outcome 1 and Outcome 2) and BMI (Outcome 6) will be assessed for a predicting relationship to Visceral Adiposity as measured by CT surface area (Outcome 4), Visceral Adiposity as measured by CT volume (Outcome 5), Framingham Cardiovascular Risk strata (Outcome 9), Liver disease (Outcome 10 and 11) or Glucose homeostasis (Outcome 12).

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Lake, MD, Principal Investigator — The University of Texas Health Science Center, Houston; John Koethe, MD, Principal Investigator — Vanderbilt University Medical Center; Jeffery Carr, DR, Principal Investigator — Vanderbilt University Medical Center
Locations (7):
- United States (7):
  - Ruane Clinical Research, Los Angeles, California
  - AIDS Healthcare Foundation, Fort Lauderdale, Florida
  - AIDS Healthcare Foundation, Miami Beach, Florida
  - Bliss Health, Orlando, Florida
  - AIDS Healthcare Foundation, New York, New York
  - Fight Community Health Centers, Philadelphia, Pennsylvania
  - Prism Health North Texas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neeland IJ, Ross R, Despres JP, Matsuzawa Y, Yamashita S, Shai I, Seidell J, Magni P, Santos RD, Arsenault B, Cuevas A, Hu FB, Griffin B, Zambon A, Barter P, Fruchart JC, Eckel RH; International Atherosclerosis Society; International Chair on Cardiometabolic Risk Working Group on Visceral Obesity. Visceral and ectopic fat, atherosclerosis, and cardiometabolic disease: a position statement. Lancet Diabetes Endocrinol. 2019 Sep;7(9):715-725. doi: 10.1016/S2213-8587(19)30084-1. Epub 2019 Jul 10. PMID 31301983
- [Background] Guilbaud L, Guedes JC, Gomez B, Gagne C, Thomas R, Szabo J. Lipohypertrophy, a preliminary estimate in the prevalence in an urban Canadian HIV clinic. Presented at the May 2019 CAHR Conference, Saskatoon SK. Poster 4420.
- [Background] Alikhani A, Morin H, Matte S, Alikhani P, Tremblay C, Durand M. Association between lipodystrophy and length of exposure to ARTs in adult HIV-1 infected patients in Montreal. BMC Infect Dis. 2019 Sep 18;19(1):820. doi: 10.1186/s12879-019-4446-9. PMID 31533648
- [Background] Koethe JR. Adipose Tissue in HIV Infection. Compr Physiol. 2017 Sep 12;7(4):1339-1357. doi: 10.1002/cphy.c160028. PMID 28915327
- [Background] Orlando G, Guaraldi G, Zona S, Carli F, Bagni P, Menozzi M, Cocchi S, Scaglioni R, Ligabue G, Raggi P. Ectopic fat is linked to prior cardiovascular events in men with HIV. J Acquir Immune Defic Syndr. 2012 Apr 15;59(5):494-7. doi: 10.1097/QAI.0b013e31824c8397. PMID 22410868
- [Background] Fourman LT, Kileel EM, Hubbard J, Holmes T, Anderson EJ, Looby SE, Fitch KV, Feldpausch MN, Torriani M, Lo J, Stanley TL, Grinspoon SK. Comparison of visceral fat measurement by dual-energy X-ray absorptiometry to computed tomography in HIV and non-HIV. Nutr Diabetes. 2019 Feb 25;9(1):6. doi: 10.1038/s41387-019-0073-1. PMID 30804324
- [Background] Lemoine M, Assoumou L, De Wit S, Girard PM, Valantin MA, Katlama C, Necsoi C, Campa P, Huefner AD, Schulze Zur Wiesch J, Rougier H, Bastard JP, Stocker H, Mauss S, Serfaty L, Ratziu V, Menu Y, Schlue J, Behrens G, Bedossa P, Capeau J, Ingiliz P, Costagliola D; ANRS-ECHAM Group. Diagnostic Accuracy of Noninvasive Markers of Steatosis, NASH, and Liver Fibrosis in HIV-Monoinfected Individuals at Risk of Nonalcoholic Fatty Liver Disease (NAFLD): Results From the ECHAM Study. J Acquir Immune Defic Syndr. 2019 Apr 1;80(4):e86-e94. doi: 10.1097/QAI.0000000000001936. PMID 30570529
- [Background] Lake JE, Stanley TL, Apovian CM, Bhasin S, Brown TT, Capeau J, Currier JS, Dube MP, Falutz J, Grinspoon SK, Guaraldi G, Martinez E, McComsey GA, Sattler FR, Erlandson KM. Practical Review of Recognition and Management of Obesity and Lipohypertrophy in Human Immunodeficiency Virus Infection. Clin Infect Dis. 2017 May 15;64(10):1422-1429. doi: 10.1093/cid/cix178. PMID 28329372
- [Background] Gabriel CL, Ye F, Fan R, Nair S, Terry JG, Carr JJ, Silver H, Baker P, Hannah L, Wanjalla C, Mashayekhi M, Bailin S, Lima M, Woodward B, Izzy M, Ferguson JF, Koethe JR. Hepatic Steatosis and Ectopic Fat Are Associated With Differences in Subcutaneous Adipose Tissue Gene Expression in People With HIV. Hepatol Commun. 2021 Feb 27;5(7):1224-1237. doi: 10.1002/hep4.1695. eCollection 2021 Jul. PMID 34278171
- [Background] Monczor AN, Li X, Palella FJ Jr, Erlandson KM, Wiley D, Kingsley LA, Post WS, Jacobson LP, Brown TT, Lake JE. Systemic Inflammation Characterizes Lack of Metabolic Health in Nonobese HIV-Infected Men. Mediators Inflamm. 2018 Sep 25;2018:5327361. doi: 10.1155/2018/5327361. eCollection 2018. PMID 30356397
- [Background] Beraldo RA, Meliscki GC, Silva BR, Navarro AM, Bollela VR, Schmidt A, Foss-Freitas MC. Comparing the Ability of Anthropometric Indicators in Identifying Metabolic Syndrome in HIV Patients. PLoS One. 2016 Feb 26;11(2):e0149905. doi: 10.1371/journal.pone.0149905. eCollection 2016. PMID 26919174
- [Background] Koethe JR, Lagathu C, Lake JE, Domingo P, Calmy A, Falutz J, Brown TT, Capeau J. HIV and antiretroviral therapy-related fat alterations. Nat Rev Dis Primers. 2020 Jun 18;6(1):48. doi: 10.1038/s41572-020-0181-1. PMID 32555389
- [Background] Pouliot MC, Despres JP, Lemieux S, Moorjani S, Bouchard C, Tremblay A, Nadeau A, Lupien PJ. Waist circumference and abdominal sagittal diameter: best simple anthropometric indexes of abdominal visceral adipose tissue accumulation and related cardiovascular risk in men and women. Am J Cardiol. 1994 Mar 1;73(7):460-8. doi: 10.1016/0002-9149(94)90676-9. PMID 8141087
- [Background] O'Neill T, Guaraldi G, Orlando G, Carli F, Garlassi E, Zona S, Despres JP, Ross R. Combined use of waist and hip circumference to identify abdominally obese HIV-infected patients at increased health risk. PLoS One. 2013 May 20;8(5):e62538. doi: 10.1371/journal.pone.0062538. Print 2013. PMID 23700409
- [Background] Hunter GR, Snyder SW, Kekes-Szabo T, Nicholson C, Berland L. Intra-abdominal adipose tissue values associated with risk of possessing elevated blood lipids and blood pressure. Obes Res. 1994 Nov;2(6):563-8. doi: 10.1002/j.1550-8528.1994.tb00106.x. PMID 16355516
- [Background] Yoo S, Sung MW, Kim H. CT-defined visceral adipose tissue thresholds for identifying metabolic complications: a cross-sectional study in the United Arab Emirates. BMJ Open. 2020 Aug 11;10(8):e031181. doi: 10.1136/bmjopen-2019-031181. PMID 32788183
- [Background] Katzmarzyk PT, Greenway FL, Heymsfield SB, Bouchard C. Clinical utility and reproducibility of visceral adipose tissue measurements derived from dual-energy X-ray absorptiometry in White and African American adults. Obesity (Silver Spring). 2013 Nov;21(11):2221-4. doi: 10.1002/oby.20519. Epub 2013 Aug 13. PMID 23794256
- [Background] Williams MJ, Hunter GR, Kekes-Szabo T, Trueth MS, Snyder S, Berland L, Blaudeau T. Intra-abdominal adipose tissue cut-points related to elevated cardiovascular risk in women. Int J Obes Relat Metab Disord. 1996 Jul;20(7):613-7. PMID 8817354
- [Background] Katzmarzyk PT, Heymsfield SB, Bouchard C. Clinical utility of visceral adipose tissue for the identification of cardiometabolic risk in white and African American adults. Am J Clin Nutr. 2013 Mar;97(3):480-6. doi: 10.3945/ajcn.112.047787. Epub 2013 Jan 30. PMID 23364010
- [Background] Lemieux S, Prud'homme D, Bouchard C, Tremblay A, Despres JP. A single threshold value of waist girth identifies normal-weight and overweight subjects with excess visceral adipose tissue. Am J Clin Nutr. 1996 Nov;64(5):685-93. doi: 10.1093/ajcn/64.5.685. PMID 8901786
- [Background] Rankinen T, Kim SY, Perusse L, Despres JP, Bouchard C. The prediction of abdominal visceral fat level from body composition and anthropometry: ROC analysis. Int J Obes Relat Metab Disord. 1999 Aug;23(8):801-9. doi: 10.1038/sj.ijo.0800929. PMID 10490780
- [Background] Falutz J, Rosenthall L, Kotler D, Zona S, Guaraldi G. Surrogate markers of visceral adipose tissue in treated HIV-infected patients: accuracy of waist circumference determination. HIV Med. 2014 Feb;15(2):98-107. doi: 10.1111/hiv.12085. Epub 2013 Sep 22. PMID 24112443
- [Background] Zhou Q, Usadel S, Kern W, Zirlik A, Mueller MC. Real world cardiovascular risk assessment using reduced DAD, SCORE and Framingham equations in a German HIV cohort. Eur Heart J. 2020;41 (Suppl. 2):ehaa946.2914.
- [Background] Beraldo RA, Meliscki GC, Silva BR, Navarro AM, Bollela VR, Schmidt A, Foss-Freitas MC. Anthropometric measures of central adiposity are highly concordant with predictors of cardiovascular disease risk in HIV patients. Am J Clin Nutr. 2018 Jun 1;107(6):883-893. doi: 10.1093/ajcn/nqy049. PMID 29868914